CLINICAL TRIAL: NCT06581848
Title: Korean Post Marketing Surveillance for ELREXFIO (Elranatamab).
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C1071029
Record Dates: First submitted 2024-08-13; First posted 2024-09-03 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Elranatamab
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elranatamab: Patients who have been prescribed Elranatamab by their physician as monotherapy for the treatment of adult patients with relapsed or refractory multiple myeloma, who have received at least three prior therapies, including a proteasome inhibitor, an immunomodulatory agent, and an anti-CD38 monoclonal antibody, and have demonstrated disease progression on the last therapy.
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — According to the approved label, the recommended doses are step-up doses of 12 mg on day 1 and 32 mg on day 4, followed by a full treatment dose of 76 mg weekly from week 2 to week 24. For patients who have received at least 24 weeks of treatment and have achieved a response, the dosing interval should transition to an every two week schedule.

SUMMARY:
This study is to assess the safety and effectiveness of Elranatamab in the real-world clinical settings for the treatment of patients with multiple myeloma in Korea.

DETAILED DESCRIPTION:
This study is an open-label, multi-center, non-comparative, observational study to assess safety and effectiveness of Elranatamab in the real-world clinical setting in patients with multiple myeloma in Korea.

During the study period within 2 years from the launch date, a whole case enrollment should be conduct according to the protocol.

The objectives of this study are to determine safety and effectiveness with Elranatamab under conditions of general clinical practice, in compliance with the regulation of the MFDS. Therefore, this study was designed according to the PMS guidelines of the MFDS.

The study population is patients who are eligible for "Indications" specified in the approved label.

All assessments described in this protocol are performed as part of normal clinical practice or standard practice guidelines for the patient population and healthcare provider specialty in the countries where this Non-interventional study (NIS) is being conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been prescribed ELREXFIO (Elranatamab) by their physician as monotherapy for the treatment of adult patients with relapsed or refractory multiple myeloma, who have received at least three prior therapies, including a proteasome inhibitor, an immunomodulatory agent, and an anti-CD38 monoclonal antibody, and have demonstrated disease progression on the last therapy.
* Patients with evidence of a personally signed and dated informed consent/assent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients with contraindication according to locally approved label of ELREXFIO (Elranatamab)
* Any patients (or a legally acceptable representative) who does not agree that Pfizer and companies working with Pfizer use his/her information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients who are eligible for "Indications" specified in the approved label.
  [INDICATIONS] Elranatamab is indicated as monotherapy for the treatment of adult patients with relapsed or refractory multiple myeloma, who have received at least three prior therapies, including a proteasome inhibitor, an immunomodulatory agent, and an anti-CD38 monoclonal antibody, and have demonstrated disease progression on the last therapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of an adverse event (AE)/ adverse drug reaction (ADR) | At least 28 days from the last dose of Elranatamab
  The safety analysis population will consist of all patients who received at least one dose of the study drug and had at least one follow-up safety evaluation.
  The numbers and proportions of patients experiencing AE and ADR will be summarized with the 95% CIs in addition to their occurrence frequencies.
Incidence of a serious AE (SAE)/ serious ADR (SADR) | At least 28 days from the last dose of Elranatamab
  The safety analysis population will consist of all patients who received at least one dose of the study drug and had at least one follow-up safety evaluation.
  The numbers and proportions of patients experiencing SAE and SADR will be summarized with the 95% CIs in addition to their occurrence frequencies.
Incidence of an unexpected AE (UAE)/ unexpected ADR (UADR) | At least 28 days from the last dose of Elranatamab
  The safety analysis population will consist of all patients who received at least one dose of the study drug and had at least one follow-up safety evaluation.
  The numbers and proportions of patients experiencing UAE and UADR will be summarized with the 95% CIs in addition to their occurrence frequencies.
Incidence of a serious unexpected AE (SUAE)/ serious unexpected ADR (SUADR) | At least 28 days from the last dose of Elranatamab
  The safety analysis population will consist of all patients who received at least one dose of the study drug and had at least one follow-up safety evaluation.
  The numbers and proportions of patients experiencing SUAE and SUADR will be summarized with the 95% CIs in addition to their occurrence frequencies.
Incidence of an adverse event special interest (AESI) | At least 28 days from the last dose of Elranatamab
  The safety analysis population will consist of all patients who received at least one dose of the study drug and had at least one follow-up safety evaluation.
  The numbers and proportions of patients experiencing AESI will be summarized with the 95% CIs in addition to their occurrence frequencies.

SECONDARY OUTCOMES:
Objective response rate (ORR) per International Myeloma Working Group (IMWG) response criteria as determined by investigator | From the first dose of the study drug until completion or discontinuation of the study or death due to any cause, whichever occurs first, assessed up to 72 months.
  The effectiveness analysis population will consist of a subset of the safety analysis population that captured at least one follow-up effectiveness assessment.
  Objective Response will encompass confirmed sCR, CR, VGPR and PR. ORR is defined as the proportion of patients with an objective response per IMWG criteria.
Progression-free survival (PFS) per IMWG response criteria as determined by investigator | From the first dose of the study drug until confirmed Progressive Disease per IMWG criteria or death due to any cause, whichever occurs first, assessed up to 72 months.
  The effectiveness analysis population will consist of a subset of the safety analysis population that captured at least one follow-up effectiveness assessment.
  PFS is defined as the time from the first dose of the study drug until confirmed PD per IMWG criteria or death due to any cause, whichever occurs first.
Time to response (TTR) per IMWG response criteria as determined by investigator | From the first dose of the study drug to the first documentation of response that is subsequently confirmed, assessed up to 72 months.
  The effectiveness analysis population will consist of a subset of the safety analysis population that captured at least one follow-up effectiveness assessment.
  TTR is defined, for patients with an objective response per IMWG criteria, as the time from the date of first dose of ELREXFIO to the first documentation of response that is subsequently confirmed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.